CLINICAL TRIAL: NCT02463162
Title: Effectiveness and Economic Impact of Advance Care Planning and Goals of Care Designations Discussions: A Randomized Controlled Trial
Brief Title: Trial of Advance Care Planning (ACP) & Goals of Care Designations (GCD) Discussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00054953
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Advance Care Planning; Goals of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This group will receive "usual care" which is to receive no intervention.
- Intervention (Experimental): This group will receive the intervention which is two Conversations Matter videos about Advance Care Planning and Goals of Care Designations respectively
  Interventions: Other: Conversations Matter videos

INTERVENTIONS:
Other: Conversations Matter videos — 2 videos about Advance Care Planning and Goals of Care Designations respectively. These 2 videos were developed by Alberta Health Services and are each 8 minutes long.
  Arms: Intervention

SUMMARY:
The Canadian population is aging and more people are living with advanced chronic diseases. At the end of life (EOL), the use of invasive medical treatments in hospitals is increasing and associated with worse outcomes. Advance Care Planning (ACP) may help improve care at EOL to be the way patients want it. ACP is a process where people think about the various options related to future health care decisions and they may communicate with a verbal or written plan of what care they would want in the EOL. Also, they may nominate a substitute decision maker if they become unable to speak for themselves. A national poll found that few Canadians have thought about or made an ACP.

Alberta Health Services has developed two videos (Videos) to help with decision making about ACP and goals of care designations(GCD). GCD are medical orders of care that (a) serve as a communication tool for HCP to assist in rapid decision making; and (b) guide HCP and patients regarding the general intent and locations of care, and interventions that are to be provided. This study will compare ACP behaviours and GCD preferences for participants who have seen the Videos with those who have not and measure the change in those behaviours and preferences at 1, 2 and 3 months. It will also look at the impact of the Videos on health care costs and service use. Participants from five patient groups (metastatic lung cancer, colorectal cancer, gynecological cancer, renal failure, and heart failure) were selected as representative of where ACP should ideally be occurring, and where data on ACP implementation is presently most lacking, and as venues in which this research is most feasible. Collecting information about patients' ACP and GCD preferences may help improve AHS decision making tools and more generally help healthcare leaders plan ways to better engage patients in the ACP process.

DETAILED DESCRIPTION:
Background: Respecting patients' preferences for treatment is a key component of high quality end of life care. Alberta Health Services (AHS) has developed tools for public, patient and healthcare provider (HCP) engagement and education (such as guidebooks, videos, and HCP training modules) to support widespread engagement in advance care planning (ACP) and determining Goals of Care Designation (GCD). However, none of these knowledge translation (KT) tools have been validated and they have not been tailored to reflect barriers in the local context.

ACP is defined as a communication process where people plan for a time when they cannot make medical decisions for themselves. It includes thinking about and communicating their preferences for future healthcare, which can include conversations with family and healthcare providers, choosing and documenting an alternate decision maker, and/or documenting preferences for healthcare for use in the event that person loses capacity for medical decision-making. These discussions can occur both informally and formally. Goals of Care Designations (GCD) are medical orders of care that (a) serve as a communication tool for HCP to assist in rapid decision making; and (b) guide HCP and patients regarding the general intent and locations of care, and interventions that are to be provided. Decisions about goals of care usually arise over time through conversations between patients, family members and the health care team.

This randomized controlled trial (RCT) will focus on the two Conversations Matter Video decision-aids developed by AHS for people and their families. The first video is an 8-minute video that describes the 5-steps of the ACP process. The second video is a 8-minute video that illustrates the resuscitative, medical and comfort levels of care outlined in the Alberta GCD policy.

Scope: This protocol relates to two of the research activities designed to evaluate the impact of ACP/GCD. The first is an RCT to evaluate the effectiveness of two videos about ACP and GCD. Participants will be recruited from settings where ACP should ideally be occurring, and where data on ACP implementation is presently most lacking. The overall aim of the RCT is to evaluate and refine these existing knowledge translation (KT) tools to optimize the quality and frequency of patient education about and engagement in ACP and determining goals of care.

The second activity measures the economic impact of the Videos in these patient populations. A significant proportion of health care resources are consumed at end of life. ACP, which emphasizes discussions, combined with GCD, may have a greater impact than advance directives alone. To be clear, the primary goal of ACP is not about cost containment, but rather, to shift a culture of care toward a patient- and family-centered approach to medical decision-making. Prospective data collection and analysis will give insight into personal and intangible costs. It will allow for relatively precise measurement of health care savings, and thereby inform health care systems on anticipated savings and prescribe shift of funding necessary for appropriate resourcing in parts of the health care system that may see increased activity because of ACP, while also improving quality of patient-centred outcomes.

Methods: The RCT will be an in-person intervention and survey at baseline, follow-up telephone survey at one month and two months, and in-person survey at three months. At baseline, researchers will assess function and ask about demographic information, quality of life, advance care planning (ACP), and goals of care (GC) preferences and goals of care designation orders (GCD). Participants will then be randomized between two arms:

1. control or "usual care"; and
2. intervention whereby participant views two videos about ACP and GCD, respectively (Videos).

Surveys will be administered by research staff. The baseline intervention and survey will take approximately 30 to 65 minutes, depending on which arm the participant is randomized to, and be collected from up to 240 participants. At one, two and three months, follow up surveys will be administered to collect data about health care services utilized, health care costs incurred, and discussions about ACP and GC with their health care providers, lawyers, financial advisors and/or clergy in the preceding month. The one and two month surveys will be approximately 10-20 minutes in length. Three-month follow-up surveys will collect data about ACP, GC preferences and GCD and will be approximately 20-40 minutes in length. Researchers will also collect data from participants' electronic medical health records about their diagnosis and co-morbidities, health services utilization and costs at 12 months prior to baseline, baseline and approximately 12 months after baseline.

Objectives:

1. Determine the effectiveness of the Videos by comparing the change from baseline to 1, 2 and 3 months of the number of participants who have had a conversation with a health care provider about ACP or GCD between two groups, namely: those who receive no intervention (usual care) and those who watch the Videos.
2. Determine the cost and economic consequences of the Videos by comparing the change from 12 months prior to baseline to and including baseline, to 1 month, 2, months, 3 months and 12 months following baseline in health care utilization and costs between the two groups described in Objective 1.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of either:

  1. heart failure classified as Class III or IV based on New York Heart Association Functional Classification or classified as Stage D based on American Heart Association/American College of Cardiology Heart Failure Classification;
  2. renal failure and on dialysis; or
  3. metastatic lung, gastrointestinal (including pancreatic) or gynecological cancer and on chemo, radiation therapy or palliative
* 19 or over
* able to communicate in English
* reside within 100 km of Edmonton or Calgary
* owns a phone

Exclusion Criteria:

* cognitive impairment which would impact ability to give informed consent
* in crisis
* first visit or in the case of renal patients, in the first month of dialysis
* participated in ACP pilot study
* visual and/or hearing impairment that would impact their ability to see and/or hear the Videos, and/or complete the assessments including the telephone follow-up interviews.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Video effectiveness measured by change from baseline in number of participants who have had a conversation with a health care provider about ACP or GCD to 1 month, 2 months and 3 months | 1 month, 2 months and 3 months
  Determine the effectiveness of the Videos by comparing the number of participants who have had a conversation with a health care provider about ACP or GCD between two groups (those who receive the intervention (usual care) and those who watch the videos
Economic impact of Videos measured by comparing change from 12 months prior to baseline in health care costs to baseline, 1 month, 2 months, 3 months and 12 months after baseline between two groups | 12 months prior to baseline, baseline, 1 month, 2 months, 3 months and 12 months after baseline
  Determine the cost and economic consequences of the Videos by comparing change in health care costs between two groups (those who receive no intervention (usual care) and those who watch the Videos)

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Fassbender, PhD, Principal Investigator — University of Alberta; Sara Davison, MD, MHSc (Bioethics), Principal Investigator — University of Alberta; Jessica Simon, MD, Principal Investigator — University of Calgary
Locations (15):
- Canada (15):
  - Peter Lougheed Centre: Heart Function Clinic, Calgary, Alberta
  - Sunridge Dialysis Unit: Hemodialysis, Calgary, Alberta
  - Southern Alberta Renal Program - Northlands Village Mall, Hemodialysis, Calgary, Alberta
  - Foothills Medical Centre: Heart Function and Heart Transplant Clinic, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Sheldon M. Chumir Health Centre: Hemodialysis, Calgary, Alberta
  - Rockyview General Hospital: Heart Function Clinic, Calgary, Alberta
  - South Calgary Health Centre: Hemodialysis, Calgary, Alberta
  - South Health Campus: Heart Function Clinic, Calgary, Alberta
  - Royal Alexandra Hospital: Renal Insufficiency Clinic and Hemodialysis Unit, Edmonton, Alberta
  - Edmonton General Continuing Care Centre: Hemodialysis, Edmonton, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Alberta Hospital: Renal Insufficiency Clinic and Hemodialysis Units, Edmonton, Alberta
  - Grey Nuns Community Hospital: Renal Insufficiency Clinic and Hemodialysis Unit, Edmonton, Alberta

REFERENCES:
- [Derived] Douglas ML, Simon J, Davison SN, Biondo P, Ghosh S, Kassam A, Fassbender K. Efficacy of Advance Care Planning Videos for Patients: A Randomized Controlled Trial in Cancer, Heart, and Kidney Failure Outpatient Settings. Med Decis Making. 2021 Apr;41(3):292-304. doi: 10.1177/0272989X20985836. Epub 2021 Jan 15. PMID 33451263